CLINICAL TRIAL: NCT06627127
Title: Multicenter Proof-of-Concept Study to Investigate the Feasibility and Respiratory Effects of Stimulating Two Functional Targets (neural And/or Muscular) for the Treatment of Obstructive Sleep Apnea
Brief Title: A Study to Investigate the Feasibility and Respiratory Effects of Stimulating Two Functional Targets (neural And/or Muscular) for the Treatment of Obstructive Sleep Apnea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Invicta Medical Inc. (Industry)
Collaborators: Adelaide Institute for Sleep Health (Other); The University of Western Australia (Other); Flinders University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IM-005
Record Dates: First submitted 2024-06-24; First posted 2024-10-04 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Sleep Apnea; Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Sleep Disorder
Keywords: Sleep Apnea device
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Wake Disorders

STUDY DESIGN:
Intervention Model Description: Multicenter, proof- of-concept (POC) study. Electrode arrays percutaneously placed under ultrasound adjacent to nerves, connected to an external pulse generator will be used to evaluate the combined effect of short-term stimulation on airflow and/or AHI.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Target stimulation (Experimental): Stimulation of the Hypoglossal nerve (HGN) or Genioglossus muscle (GG) and a second functional target (Ansa Cervicalis - AC) or the strap muscles (sternohyoid and sternothyroid).
  Interventions: Device: Target stimulation (HGN, AC, GG, Strap muscles)

INTERVENTIONS:
Device: Target stimulation (HGN, AC, GG, Strap muscles) — Stimulation of the HGN or GG along with AC or strap muscles.

SUMMARY:
This proof-of-concept study is to collect acute and short-term sub-acute (if applicable) changes in respiratory parameters following the percutaneous placement of electrode arrays. Acute placement and data collection will be conducted while performing a Drug Induced Sleep Endoscopy (DISE) where the goal will be to quantify changes in airflow with stimulation. Data will also be collected during a one- or two-night polysomnography (PSG) to investigate airflow and sleep stability responses with and without different levels of stimulation during sleep. Where feasible, OSA severity data will be collected, as measured via the apnea/hypopnea index (AHI) with stimulation versus without stimulation as a secondary objective. Both data collections will be done when stimulating the hypoglossal nerve (HGN) or Genioglossus muscle (GG) and a second functional target (Ansa Cervicalis - AC) or the strap muscles (sternohyoid and sternothyroid) with a set of electrode arrays either in combination or separately.

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following inclusion criteria to be eligible for inclusion in this study:

* Age above 18 years not under guardianship, under curatorship or under judicial protection.
* Body Mass Index (BMI) < 35 kg/m2.
* OSA (15 < AHI < 80 events/h sleep) documented by a sleep study performed during the past 24 months in the absence of any major weight change or other medical issues.
* Subject must be eligible for a diagnostic DISE or surgical procedure (acute study measures only).
* Written informed consent obtained from the subject prior to performing any study specific procedure.
* Willing and capable to comply with all study requirements, including specific lifestyle considerations, evaluation procedures and questionnaires for the whole duration of the trial.

Exclusion Criteria:

Subjects meeting any of the following criteria will be excluded from participation in this study:

* Major anatomical or functional abnormalities that would impair the ability of the electrode arrays to be positioned.
* Significant comorbidities that contraindicate surgery or general anesthesia/DISE
* Significant tongue weakness
* Any other chronic medical illness or condition that contraindicates a surgical procedure or general anesthesia/DISE in the judgment of the investigator.
* Prior surgery or treatments that could compromise the placement and effectiveness of the electrode array systems:

  * Airway cancer surgery or radiation,
  * Mandible or maxilla surgery in the previous 3 years (not counting dental treatments),
* Other upper airway surgery to remove obstructions related to OSA in the previous 3 months (e.g., uvulopalatopharyngoplasty (UPPP), tonsillectomy, nasal airway surgery),
* Prior hypoglossal nerve stimulation device implantation.
* Currently pregnant, or breastfeeding during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Feasibility of technical delivery in stimulating target nerves or muscles | Day 0 to 3
  Assessment of the technical ability to simulate the target nerves and/or muscles as observed during nasoendoscopy and ultrasound imaging
Assessment of the required stimulation amplitude | Day 0 to 3
  Assess the required stimulation amplitude measured in milliamps (mA) to improve airflow during stimulation as assessed by direct visualisation of the amplitude.
Feasibility of participant recruitment and retention | Day 0 to 30
  Demonstration of participant recruitment and retention rates for a POC target stimulation in OSA participant study, measured by direct participant recruitment numbers and during on study.

SECONDARY OUTCOMES:
Acute increase in airflow measured during target stimulation | Day 0 to 3
  Demonstration of acute increase in airflow when stimulating the HGN or GG in combination with the AC or strap muscles during a flow limited event (hypopnea or apnea), measured in liters per second (L/s) using pneumotachometer.
Assessment of acute airway opening during target stimulation | Day 0 to 3
  Demonstration of changes in acute cross-sectional airway opening measured under nasoendoscopy when stimulating two functional targets simultaneously (i.e., the HGN and AC). Video imaging and physician interpretation of nasoendoscopic images will be used to review outcome measures.
Assessment of sub-acute airflow increase and/or AHI reduction during target stimulation during a sleep study. | Day 0 to 3
  Demonstration of in sub-acute flow increase and/or AHI reduction when stimulating two functional targets simultaneously during sleep as measured with polysomnography (PSG), measured in liters per second (L/s) using pneumotachometer.

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Illawara ENT, Wollongong, New South Wales
  - Complete ENT, Brisbane, Queensland
  - Adelaide Institute for Sleep Health, Flinders University, Adelaide, South Australia
  - Perth Head and Neck Surgery, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No